CLINICAL TRIAL: NCT04540302
Title: Prospective, Randomized, Controlled, Multicenter Study Comparing the Merit WRAPSODY™ Endovascular Stent Graft to Percutaneous Transluminal Angioplasty for Treatment of Venous Outflow Circuit Stenosis or Occlusion in Hemodialysis Patients. The WAVE Study
Brief Title: The Merit WRAPSODY AV Access Efficacy Study (WAVE)
Acronym: WAVE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Merit Medical Systems, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CVO-P3-20-01
Record Dates: First submitted 2020-09-01; First posted 2020-09-07 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-04

CONDITIONS: Venous Stenosis; Venous Occlusion
Keywords: AVF; AVG; AV fistula; AV graft
MeSH Terms: conditions — Arteriovenous Fistula

STUDY DESIGN:
Intervention Model Description: The study comprises 2 independent cohorts:
  1. Up to 244 AVF Peripheral Subjects (1:1 randomization, with approximately 122 in the study treatment and control groups)
  2. Up to 113 AVG Anastomosis Subjects (no randomization, comparison to Performance Goals)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (3):
- AVF Peripheral study treatment group (Experimental): Subjects randomised to treatment with the WRAPSODY Endovascular Stent Graft
  Interventions: Device: Merit WRAPSODY Endovascular Stent Graft
- AVF Peripheral control group (Other): Subjects randomised to treatment with standard percutaneous transluminal angioplasty (PTA)
  Interventions: Device: PTA
- AVG Anastomosis (Experimental): All subjects in this single arm cohort will receive treatment with the WRAPSODY Endovascular Stent Graft
  Interventions: Device: Merit WRAPSODY Endovascular Stent Graft

INTERVENTIONS:
Device: Merit WRAPSODY Endovascular Stent Graft — Target lesion treated with stent graft placement
  Arms: AVF Peripheral study treatment group; AVG Anastomosis
Device: PTA — Target lesion treated with standard percutaneous transluminal angioplasty (PTA)
  Arms: AVF Peripheral control group

SUMMARY:
The purpose of the study is to demonstrate the safety and efficacy of the Merit WRAPSODY Endovascular Stent Graft for treatment of stenosis or occlusion within the dialysis access outflow circuit

ELIGIBILITY:
Inclusion Criteria:

* Subject provides written informed consent
* Subject is male or female, with an age ≥ 18 years at date of enrollment.
* Subject is willing to undergo all follow-up assessments.
* Subject has a life expectancy ≥ 12 months.
* Subject is undergoing chronic hemodialysis.
* Subject has either a mature AVF or AVG in the arm.
* Target lesion(s) involves a de novo stenotic or non-stented restenotic lesion.
* Target lesion has ≥50% stenosis.
* Target lesion(s) reference vessel diameter is between 5.0 mm and 14.0 mm

Exclusion Criteria:

* Subject has a known or suspected infection of the hemodialysis access site, systemic infection and/or septicemia.
* Subject has a stroke diagnosis within 3 months prior to enrollment.
* Subject has a history of unstable angina or myocardial infarction within 60 days prior to enrollment.
* Subject is pregnant, breastfeeding, or intending to become pregnant within the next year.
* Target lesion is located within a stent / stent graft.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 357 (Estimated)
Dates: Start 2021-03-09 (Actual); Primary Completion 2024-02-22 (Actual); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects without any localized or systemic safety events (Primary Safety Endpoint) | 30 days
  Proportion of subjects without any localized or systemic safety events through 30 days post-index procedure that affect the access or venous outflow circuit and resulted in reintervention, hospitalization, or death (not including stenosis or thrombosis). Endovascular procedures performed to treat safety events after the index study procedure will be considered surgeries.
Proportion of subjects with Target Lesion Primary Patency (TLPP) (Primary Effectiveness Endpoint:) | 6 months
  Proportion of subjects with Target Lesion Primary Patency (TLPP) at 6 Months. TLPP is defined as freedom from clinically-driven target lesion revascularization (CD-TLR) or target lesion thrombosis measured through 6 months post-procedure, which is the time interval of uninterrupted patency after study procedure to the next intervention performed on the target lesion or uncorrectable target lesion occlusion.

SECONDARY OUTCOMES:
Proportion of subjects with Target Lesion Primary Patency | 12 and 24 months
Proportion of subjects with Assisted Target Lesion Primary Patency (aTLPP) | 6, 12 and 24 months
Proportion of subjects with Access Circuit Primary Patency (ACPP) | 6, 12 and 24 months
Proportion of subjects with Post-Procedure Secondary Patency | 6, 12 and 24 months
Rates of procedure- and device-related adverse events involving the access circuit | Index procedure, 30 days, and months 6, 12 and 24.

CONTACTS AND LOCATIONS:
Overall Officials: Mahmood K Razavi, MD, Principal Investigator — St. Joseph's Hospital, Orange, CA; Robert Jones, MD, Principal Investigator — The Queen Elizabeth Hospital
Locations (43):
- United States (33):
  - Southwest Kidney institute (SKI) Vascular Center, Tempe, Arizona
  - Pima Heart and Vascular, Tucson, Arizona
  - St. Joseph Hospital, Orange, California
  - Vascular Care Connecticut, Darien, Connecticut
  - Nephrology Associates, Newark, Delaware
  - First Coast Cardiovascular Institute, Jacksonville, Florida
  - Open Access Miami, LLC, Miami, Florida
  - Leesburg Vascular Access Center & Discovery Medical Research, Oscala, Florida
  - Coastal Vascular and Interventional, Pensacola, Florida
  - Chicago Access Center, Chicago, Illinois
  - Northwestern Medical Center, Chicago, Illinois
  - Indiana University Hospital and Methodist Hospital, Indianapolis, Indiana
  - King's Daughters Medical Center, Ashland, Kentucky
  - Brigham and Women's Faulkner Hospital, West Roxbury, Massachusetts
  - Michigan Vascular Access Center, Flint, Michigan
  - Vascular Institute of Atlantic Medical Imaging, Vineland, New Jersey
  - UNC Health, Chapel Hill, North Carolina
  - Charlotte Radiology, Charlotte, North Carolina
  - NC Heart and Vascular Research, Raleigh, North Carolina
  - North Carolina Nephrology Raleigh Access, Raleigh, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - University Pittsburg Medical Center, Pittsburgh, Pennsylvania
  - Providence Access Center, Providence, Rhode Island
  - Prisma Health System Upstate, Greenville, South Carolina
  - Soltero Cardiovascular Research Center, Dallas, Texas
  - Renal Disease Research Institute, Dallas, Texas
  - PPG Health PA, DBA-Tarrant Vascular, Fort Worth, Texas
  - Global Kidney Associates, Houston, Texas
  - Houston Methodist Hospital, Houston, Texas
  - University of Texas Health - Memorial Hermann Katy Hospital, Katy, Texas
  - CDVA, Pasadena, Texas
  - Dallas Nephrology Associates, Plano, Texas
  - Sentara Vascular Specialists, Virginia Beach, Virginia
- Brazil (4):
  - Instituto Santa Marta De Ensino E Pesquisa, Brasília
  - Real Hospital Português de Beneficência em Pernambuco, Recife
  - Hospital Universitário Pedro Ernesto, Rio de Janeiro
  - Instituto Dante Pazzanese de Cardiologia, São Paulo
- Toronto General Hospital, Toronto, Canada
- United Kingdom (5):
  - Queen Elizabeth Hospital, Birmingham
  - Dorset County Hospital, Dorchester
  - Royal London Hospital, London
  - Churchill Hospital, Oxford
  - Lister Hospital, Stevenage